CLINICAL TRIAL: NCT03404791
Title: A Multicenter Study Evaluating Safety and Efficacy of TAR-200 in Subjects With Muscle-Invasive Urothelial Carcinoma of the Bladder Who Are Ineligible for or Refuse Cisplatin-based Chemotherapy and Who Are Unfit for Radical Cystectomy
Brief Title: A Study of TAR-200 in Participants With Muscle-Invasive Urothelial Carcinoma of the Bladder Who Are Ineligible for or Refuse Cisplatin-based Chemotherapy and Who Are Unfit for Radical Cystectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108889; TAR-200-103 (Other: Janssen Research & Development, LLC); 2017-003107-21 (EudraCT Number); NCT04559594 (obsolete NCT alias)
Record Dates: First submitted 2017-12-28; First posted 2018-01-19 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants Ineligible for Radical Cystectomy (Experimental): Participants will receive the TAR-200 transuretherally on Day 0 in to the bladder through an Inserter and gradually releases gemcitabine during the 21-day indwelling period before being removed on Day 21 via flexible or rigid cystoscopy. Participants will undergo an 84-day induction period comprised of four consecutive 21-day dosing cycles. Participants may undergo 21 day cycle every 3 months for a maximum of 3 cycles as maintenance (Up to 14 months). Each TAR-200 system will be removed at 21 days after insertion.
  Interventions: Drug: TAR-200

INTERVENTIONS:
Drug: TAR-200 — TAR-200 will be placed for 21-day dosing cycles, with up to 7 doses per participant.
  Other Names: Gemcitabine-Releasing Intravesical System (GemRIS)

SUMMARY:
The purpose of this study is to evaluate both the safety and tolerability of up to 4 dosing cycles of TAR-200 for 21 days per dosing cycle in the induction period.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of non-metastatic muscle-invasive urothelial cell carcinoma of the bladder
* Participant must have been as fully resected as possible per the physician's judgment
* Participants must be deemed unfit for RC due to comorbid conditions with a risk of mortality
* Participants must refuse or be deemed ineligible for cisplatin-based chemotherapy
* Participant must refuse or not be eligible for radiotherapy

Exclusion Criteria:

* Other active malignancies
* Presence of any bladder or urethral anatomic feature that in the opinion of the Investigator may prevent the safe placement, indwelling use, or removal of TAR-200
* Pyeloureteral tube externalized to the skin (ureteral stent or unilateral nephrostomy tube is allowed)
* Evidence of bladder perforation during diagnostic cystoscopy
* Concurrent clinically significant infections as determined by the treating Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to Day 84
  An Adverse Event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study.

SECONDARY OUTCOMES:
Percentage of Participants with Clinical Complete Response (cCR) | Up to Day 360
  Percentage of Participants with Clinical Complete Response (cCR) will be reported as assessed by cystoscopy, pelvic computed tomography (CT), magnetic resonance imaging (MRI), positron emission tomography (PET), and biopsy (at 12 weeks only, unless clinically indicated).
Percentage of Participants with Clinical Partial Response (cPR) | Up to Day 360
  Percentage of participants with clinical partial response (cPR) will be reported as assessed by cystoscopy, pelvic computed tomography (CT), magnetic resonance imaging (MRI), positron emission tomography (PET), and biopsy (at 12 weeks only, unless clinically indicated).
Percentage of Participants with Stable Disease (SD) | Up to Day 360
  Percentage of participants with stable disease (SD) will be reported as assessed by cystoscopy, pelvic computed tomography (CT), magnetic resonance imaging (MRI), positron emission tomography (PET), and biopsy (at 12 weeks only, unless clinically indicated).
Percentage of Participants with Disease Progression | Up to Day 360
  Percentage of participants with disease progression as assessed by cystoscopy, pelvic computed tomography (CT), magnetic resonance imaging (MRI), positron emission tomography (PET), and biopsy (at 12 weeks only, unless clinically indicated)
Symptom Control | Up to Day 360
  Symptom Control is defined as changes in bladder-related symptoms per the protocol-specified bladder symptom (Urinary frequency, Nocturia, Hematuria and Dysuria/pain) and toxicity grading system (Grade 0-3).
Time to Intervention for Symptom Control | Up to Day 360
  Time to intervention for symptom control, defined as the time from the date of the first TAR-200 insertion to the date of intervention for symptom palliation.
Time to Progression | Up to Day 360
  Time to progression, defined as the time from the date of the first TAR-200 insertion to the date of first occurrence of progression.
Percentage of Participants Undergoing Post-treatment Interventions by 3, 6, 9, and 12 Months | Up to 3, 6, 9, and 12 Months
  Percentage of participants undergoing post-treatment interventions for the management of local symptoms by 3, 6, 9, and 12 months.
Percentage of Participants Surviving at 12, 24, and 36 Months | At 12, 24, and 36 months
  Percentage of participants surviving at 12, 24, and 36 months compared to all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (12):
- United States (9):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - North Georgia Urology Center, Dalton, Georgia
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Michigan Institute of Urology, Troy, Michigan
  - University of Rochester, Rochester, New York
  - Urology Associates, PC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - North Austin Urology, Austin, Texas
  - Urology of Virginia, PLCC, Virginia Beach, Virginia
- Spain (3):
  - Fund. Puigvert, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Inst. Valenciano de Oncologia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency